CLINICAL TRIAL: NCT06586281
Title: Elucidating Shared Mechanisms Contributing to Non-Alcoholic Fatty Liver Disease (NAFLD) and Psoriatic Arthritis (PsA) Disease Severity With Guselkumab Therapy
Brief Title: Elucidating Shared Mechanisms Contributing to NAFLD and PsA Disease Severity With Guselkumab Therapy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Diego (Other)
Collaborators: Janssen Scientific Affairs, LLC (Industry)
Responsible Party: Principal Investigator, Monica Guma, Professor, University of California, San Diego
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 809662
Record Dates: First submitted 2024-08-29; First posted 2024-09-19 (Actual); Last update posted 2025-04-03 (Actual); Status verified 2025-03

CONDITIONS: Psoriatic Arthritis
MeSH Terms: conditions — Arthritis, Psoriatic | interventions — guselkumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- psoriatic arthritis patients (Experimental): Adults with active PsA and diagnosed NAFLD
  Interventions: Drug: Guselkumab

INTERVENTIONS:
Drug: Guselkumab — This is a longitudinal study consisting of a two-time visit by psoriatic arthritis patients. The aim of the study is to determine the effect of biological therapies in liver disorders in patients with psoriatic arthritis.
  Other Names: Tremfya

SUMMARY:
While many studies examine Nonalcoholic fatty liver disease (NAFLD), little is known about its progression to high-risk nonalcoholic steatohepatitis (NASH) in PsA patients. Shared disease mechanisms may explain the increased severity in PsA. This study involves two visits from PsA patients with NAFLD and active disease signs (e.g., swollen joint, enthesitis, or psoriatic plaque). It aims to assess the impact of biological therapies on liver disorders, joints, and skin in PsA patients.

DETAILED DESCRIPTION:
Nonalcoholic fatty liver disease (NAFLD), ranging from benign steatosis to severe nonalcoholic steatohepatitis (NASH), is increasingly common and linked to cirrhosis. Patients with psoriatic arthritis (PsA) are at higher risk for NAFLD and NASH, partly due to methotrexate (MTX) use, which is associated with hepatotoxicity. Key cytokines involved in PsA, such as TNF, IL-17, and IL-23, may also contribute to NAFLD progression.

The proposed study aims to explore shared pathogenic pathways in NAFLD and PsA by evaluating the role of IL-17/23 through imaging, metabolomics, and synovial biopsies. Ultrasound-guided synovial biopsy, a safe and effective method, will be used to obtain tissue samples, enabling the identification of new molecular signatures and therapeutic targets to improve treatment of joint diseases.

ELIGIBILITY:
Inclusion Criteria:

1. Adults with diagnosis of PsA fulfilling the classification for PsA (CASPAR) criteria.
2. Must have:

1 or more swollen joint(s) and/or one or more active sites of enthesitis

3. AND/OR

1 or more psoriatic plaques

4. No changes in the regular medication regimen within the last three months, and no use of systemic and/or chronic steroids within 8 weeks leading up to the study.

5. Overweight or obese by BMI ≥ 25.0 kg/m2 or ≥ 23.0 for Asian participants

6. Patients are starting Guselkumab therapy for PsA as indicated by primary rheumatologist

7. Elevated liver fat on controlled attenuation parameter (CAP) ≥ 288 dB/m, which is consistent with NAFLD after exclusion of secondary causes of liver disease.

Exclusion Criteria:

1. Patients with prior exposure to IL12/23i, IL-17i, JAKi, or TYK2i. Patients with exposure to more than 2 TNFi.
2. Evidence of other causes of chronic liver disease

   * Hepatitis B as defined as presence of hepatitis B surface antigen (HBsAg).
   * Previous or current infection with Hepatitis C as defined by presence of hepatitis C virus Abin serum (anti-HCV Ab).
   * Autoimmune hepatitis as defined by anti-nuclear antibody (ANA) of 1:160 or greater and liver histology consistent with autoimmune hepatitis or previous response to immunosuppressive therapy.
   * Autoimmune cholestatic liver disorders as defined by elevation of alkaline phosphatase and anti-mitochondrial antibody of greater than 1:80 or liver histology consistent with primary biliary cirrhosis or elevation of alkaline phosphatase and liver histology consistent with sclerosing cholangitis.
   * Wilson disease as defined by ceruloplasmin below the limits of normal and liver histology consistent with Wilson disease.
   * Alpha-1-antitrypsin deficiency as defined by alpha-1-antitrypsin level less than normal and liver histology consistent with alpha-1-antitrypsin deficiency.
   * Hemochromatosis as defined by presence of 3+ or 4+ stainable iron on liver biopsy and homozygosity for C282Y or compound heterozygosity for C282Y/H63D.
   * Drug-induced liver disease as defined on the basis of typical exposure and history.
   * Bile duct obstruction as shown by imaging studies.
   * History of gastrointestinal bypass surgery or ingestion of medications known to produce steatosis, such as corticosteroids, high-dose estrogen, tamoxifen, amiodarone or tetracycline in the previous 6 months.
   * Evidence of cirrhosis or previously known cirrhosis based on the results from previous liver biopsy or history of portal hypertension presented by ascites, hepatic encephalopathy or varices
   * Presence of regular and/or excessive use of alcohol (defined as >30g/day for males and >15g/day for females) for a period longer than 2 years at any times in the last 10 years
   * Serum creatinine > 2.0 mg/dL
   * The subject is a pregnant or nursing female or is planning to become pregnant
   * Life expectancy less than 5 years
3. History of known HIV infection

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-06-01 (Estimated); Primary Completion 2026-09-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Change in NAFLD severity | 24 weeks
  Defined by MRI-PDFF responders (relative change in liver fat ≥30%) vs non-responders (relative change in liver fat <30%) at Week 24.

SECONDARY OUTCOMES:
Change from baseline in skin psoriasis severity | 24 weeks
  Defined by PASI90 (Psoriasis Area and Severity Index) response in patients with plaque psoriasis at baseline
Change in joint arthritis | 24 weeks
  Defined by change of 7.25 of DAPSA (Disease activity in Psoriatic Arthritis) from baseline in patients with at least 1 swollen joint at baseline.
Change in ALT Levels | 24 weeks
  Defined by at least 17 U/L in patients with elevated ALT at baseline (defined as ≥30 U/L).

CONTACTS AND LOCATIONS:
Locations (1):
- University of California, San Diego, San Diego, California, United States

IPD SHARING:
Plan to Share IPD: No